CLINICAL TRIAL: NCT05977478
Title: Characterization of Tissue Biochemical Composition in Gastric Precancerous/Cancerous Lesions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Collaborators: Endofotonics Pte Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022/00489
Record Dates: First submitted 2023-07-07; First posted 2023-08-04 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-06

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SPECTRA IMDx™. (Experimental): During endoscopy, the endoscopist will first locate the precancerous/cancerous gastric lesions using HD-WLE. Upon location of the lesion, the endoscopist will use the SPECTRA IMDx™ probe to capture the Raman spectra from the lesion and its adjacent normal mucosa.
  Interventions: Device: SPECTRA IMDx™

INTERVENTIONS:
Device: SPECTRA IMDx™ — In this study, SPECTRA IMDxTM system will be used to capture the Raman spectra to correlate to histopathology results and mass spectrometry profiling results.

SUMMARY:
This is a study intended to utilize endoscopic biopsies from gastric precancerous/ cancerous lesions and adjacent normal mucosa to characterize tissue biochemical composition changes as determined by mass spectrometry lipidomic/ proteomic profiling, and correlate these changes with histopathologic results, and Raman spectra as determined by SPECTRA IMDx™. The study site will be National University Hospital.

DETAILED DESCRIPTION:
This is a study intended to utilize endoscopic biopsies from gastric precancerous/ cancerous lesions and adjacent normal mucosa to characterize tissue biochemical composition changes as determined by mass spectrometry lipidomic/ proteomic profiling, and correlate these changes with histopathologic results, and Raman spectra as determined by SPECTRA IMDx™. The study site will be National University Hospital. Subjects will be patients with current or known history of gastric dysplasia and gastric cancer, or endoscopic surveillance after previous endoscopic or surgical resection for gastric dysplasia or gastric cancer, for which upper gastrointestinal endoscopy is indicated. Patients who meet the study criteria and have consented to participate in the study will undergo upper gastrointestinal endoscopy examination as per standard practice.

During endoscopy, the endoscopist will first locate the precancerous/cancerous lesions using HD-WLE. Upon location of the lesion, the endoscopist will use the SPECTRA IMDx™ probe to capture the Raman spectra from the lesion and its adjacent normal mucosa. Two biopsies will be obtained from the lesion, and two biopsies from adjacent normal mucosa at the exact sites where the SPECTRA IMDx probe has been placed. One biopsy each from the lesion and from normal mucosa will be sent for histopathologic examination. Another biopsy each from the lesion and normal mucosa will be snap-freeze, stored in liquid nitrogen immediately, and transferred to mass spectrometry service provider for lipidomic and proteomic profiling. Histopathology results and mass spectrometry profiling results will be correlated to Raman spectra. Subjects will receive the standard care assessments throughout the study according to the hospital's standard procedures. No follow-up is needed in this study.

ELIGIBILITY:
Inclusion Criteria:

1. They are aged 21 years and above
2. They will be undergoing upper gastrointestinal endoscopy for any of the following:

   1. Current or known history of gastric dysplasia and gastric cancer, or
   2. Endoscopic surveillance after previous endoscopic or surgical resection for gastric dysplasia or gastric cancer.
3. They must be mentally competent.
4. They must be willing and able to comply with all study procedures.

Exclusion Criteria:

1. Subjects with bleeding disorders, such as haemophilia, in whom biopsies are contraindicated.
2. Subjects with active bleeding or coagulopathy precluding biopsies.
3. Pregnant subjects.
4. The subject with severe co-morbid illness, such as end-stage renal failure (ESRF), congestive cardiac failure (CCF) and advanced liver cirrhosis.
5. Subjects with other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may interfere with the interpretation of study results or would make the subject unsuitable for entry into the study

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2022-10-27 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Correlating tissue biochemical composition with the Raman spectra and histopathologic results to differentiate between the gastric disease states based on distinct features in the biochemical composition of pre-cancerous / cancerous lesions. | 18 moths
  To utilize endoscopic biopsies from gastric precancerous/ cancerous lesions and adjacent normal mucosa to characterize tissue biochemical composition changes as determined by mass spectrometry lipidomic/ proteomic profiling, and correlate these changes with histopathologic results, and Raman spectra as determined by SPECTRA IMDx™.

CONTACTS AND LOCATIONS:
Overall Officials: Guowei Kim, MBBS, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No